CLINICAL TRIAL: NCT04971980
Title: A Phase 1/2a, Open-Label Study to Evaluate the Safety and Efficacy of a Single Intravenous Infusion of BC-U001, a Human Umbilical Cord-Derived Mesenchymal Stem Cell Product, for Rheumatoid Arthritis
Brief Title: Safety and Efficacy Study of Human Umbilical Cord-Derived Mesenchymal Stem Cells(BC-U001) for Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Baylx Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BC-U001-RA2019
Record Dates: First submitted 2021-06-30; First posted 2021-07-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis
Keywords: mesenchymal stem cell; autoimmune disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hUC-MSC infusion (BC-U001) (Experimental): Cohort 1: Low-dose BC-U001 Cohort 2: Medium-dose BC-U001 Cohort 3: High-dose BC-U001
  Interventions: Drug: hUC-MSC infusion (BC-U001)

INTERVENTIONS:
Drug: hUC-MSC infusion (BC-U001) — The participants are intravenously administered a single infusion of hUC-MSC at 0.5x10^6 cells/kg body weight, 1.0x10^6 cells/kg body weight, 1.5x10^6 cells/kg body weight for low-dose cohort, medium-dose cohort and high-dose cohort respectively.

SUMMARY:
BC-U001 is an allogeneic fresh human umbilical cord-derived mesenchymal stem cell product, which showed therapeutic potential for rheumatoid arthritis(RA) based on its anti-inflammatory, immunomodulatory and tissue repair activities. The primary objective of this open-label, non-randomized, dose-escalation study is to evaluate the safety and tolerability of a single intravenous infusion of BC-U001 for RA patients using a 3+3 design.

DETAILED DESCRIPTION:
This study will enroll RA patients who still remained moderate-to-high disease activity after conventional synthetic DMARDs (csDMARDs) therapy. All participants are informed about the study procedures and potential risks and are required to provide written informed consent prior to study begin.

A 3+3 dose escalation design will be implemented. Three ascending dose cohorts (3 participants/cohort) will be treated successively to identify the maxium tolerated dose (MTD) and/or a recommended dose for phase II study. Dose escalation will be terminated if the dose-limiting toxicities (DLT) are observed in 2 participants during the 28-day follow-up within cohort.

DLT was defined as any ≥grade 3 non-hematological toxicity or grade 4 hemtological toxicity according to CTCAE v5.0, which was related to the investigational product determined by investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 (inclusive)
2. Patients who are diagnosed with rheumatoid arthritis following the 2010 ACR/EULAR classification criteria
3. Patients who still remain moderate-to-high disease activity, i.e. DAS28>3.2 at screening and study baseline, after standard csDMARDs therapy
4. Patients who are positive for rheumatoid factors (RF) and/or anti-CCP antibody
5. Patients who are clinically stable with no significant changes in physical condition from screening to study baseline
6. Patients who are available and willing to comply with all study procedures
7. Patients must be informed of the investigational nature of this study and give written informed consent in accordance with the institutional and hospital guidelines

Exclusion Criteria:

1. Infections of hepatitis B, hepatitis C, active or latent tuberculosis, or positive for human immunodeficiency virus (HIV)1 or HIV2
2. Any history of ongoing, significant infections or recent serious infection, i.e., requiring hospitalization and or IV antimicrobial treatment in the 3 months prior to screening
3. Any active inflammatory diseases other than RA
4. Serum aminotransferase (ALT or AST) levels ≥ 2x upper limits of normal
5. Creatinine clearance rate (Ccr) < 45 ml/min calculated by Cockcroft-Gault formula
6. Severe chronic obstructive pulmonary disease or known lung disease except for mild asthma treated with bronchodilators
7. Any coexistent active major medical diagnosis of clinically significant cardiovascular, neurological psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease), or hematological abnormalities that are likely to interfere with patient compliance or study assessments/procedures in the investigators' opinion
8. History of cerebrovascular accident (stroke) within 1 year before screening
9. Clinically significant heart disease (New York Heart Association, class III and class IV)
10. Surgery or trauma (e.g. contusions, abrasions, stab wounds, cutting wounds, crush injuries, impact injuries, and firearm injuries etc.) within 14 days before enrollment that are not approporiate to participate in study in investigators' opinion
11. Pregnant, breastfeeding, or desire to become pregnant or unwilling to practice birth control during participation in the study and for twelve months after completing the study infusion, unless surgically sterilized or postmenopausal during the study
12. Corticosteroid usage at a high dose (i.e., IV or IM corticosteroids or use of oral prednisone equivalent >10 mg/day) or not at a stable dose for the treatment of RA or other diseases within 28 days prior to randomization.
13. Known allergies or had a history of allergy to minor molecular heparinum and human serum albumin that are likely to interfere with patient compliance or study assessments/procedures in the investigators' opinion
14. Already participating in another interventional clinical trial or participated in another interventional clinical trial within 3 months before screening
15. Clinical history of malignancy with the exception of adequately treated cervical carcinoma in situ or basal cell carcinomas
16. Other situations that are not approporiate to participate in study in investigators' opinion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number and frequency of adverse events (AEs) | Up to day 28±3
  Adverse events are assessed by CTCAE 5.0 up to 28±3 days. The flexible change of ±3 days is set for the convenience of patients. Day 1 refers to the day the participant accept BC-U001 infusion.
Changes of vital signs from 1 hour after infusion to day 28±3 | Up to day 28±3
Changes of complete blood count (CBC) from day 1 to day 28±3 | Up to day 28±3
Changes of blood biochemical from day 1 to day 28±3 | Up to day 28±3
Changes of coagulation function from day 1 to day 28±3 | Up to day 28±3
Routine urine analysis | Up to day 28±3
Urine pregnancy test (female only) | 28±3 days
Cardiac rate measured by twelve-lead electrocardiogram | Up to day 28±3

SECONDARY OUTCOMES:
Percentage of participants achieving ACR20 | Up to day 28±3
Percentage of participants achieving ACR50 | Up to day 28±3
Percentage of participants achieving ACR70 | Up to day 28±3
Change from baseline of the disease activity score based on DAS28-CRP | Up to day 28±3
Change from baseline of the disease activity score based on DAS28-ESR | Up to day 28±3
EULAR response | Up to day 28±3
Change from baseline of the health assessment questionnaire(HAQ) score | Up to day 28±3
Change from baseline of the simplified disease activity index (SDAI) score | Up to day 28±3
Change from baseline of the clinical disease activity index (CDAI) score | Up to day 28±3
Change from baseline of TNF-α level | Up to day 28±3
Change from baseline of IL-6 level | Up to day 28±3

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, M.D., Ph.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital (Dongdan campus), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No